CLINICAL TRIAL: NCT05366712
Title: Nexus Evaluation Primary Trident II UNcemented shEll (NEPTUNE): A Longitudinal Cohort Study of the Hydroxyapatite Coated Trident II Acetabular System in Total Hip Arthroplasty
Brief Title: Nexus Evaluation Primary Trident II Uncemented Shell
Acronym: NEPTUNE
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: NHS Lothian (Other Government)
Collaborators: University of Edinburgh (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AC20120
Record Dates: First submitted 2022-05-04; First posted 2022-05-09 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: Arthritis of Hip; Hip Dysplasia; Hip Arthropathy; Hip Osteoarthritis
Keywords: Arthroplasty; Uncemented; Hip; Trident II
MeSH Terms: conditions — Hip Dislocation; Osteoarthritis, Hip

STUDY DESIGN:
Intervention Model Description: Prospective Cohort Study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Trident® II HA coated shells (Experimental): Patients will receive a Trident® II acetabular component as part of primary total hip arthroplasty at the study centre. This component is CE marked and widely available for use by UK surgeons. The Trident® II shells are HA coated, cementless, press-fit acetabular shells composed of a Titanium (Ti-6Al-4V) substrate featuring a CpTi roughened surface with PureFix™ HA.
  Interventions: Device: Stryker Trident® II HA coated cementless acetabula component

INTERVENTIONS:
Device: Stryker Trident® II HA coated cementless acetabula component — New acetabula component.

SUMMARY:
This is a prospective cohort study assessing the survival of a new acetabula component which is based on the original Trident acetabular system (cementless shell) which is used for Total Hip Arthroplasty. The manufacturer recently introduced the evolution of this product, the Trident® II acetabular shell which was launched in 2017. This implant is CE marked and is now widely available for the UK market, however has minimal clinical outcomes data to support its use. As part of a stepwise introduction of devices to orthopaedic practice. This study will report the 10 year implant survival and patient functional outcomes of this new implant.

DETAILED DESCRIPTION:
125 patients will be recruited at a single-centre as part of a, phase-4 post-market surveillance, prospective cohort study

This is a 10-year study of the Trident II acetabular component as part of total hip replacement at the Royal Infirmary of Edinburgh, NHS Lothian.

Patients will receive a Trident® II acetabular component as part of primary total hip arthroplasty at the study centre. This component is CE marked and widely available for use by UK surgeons. The Trident® II shells are HA coated, cementless, press-fit acetabular shells composed of a Titanium (Ti-6Al-4V) substrate featuring a CpTi roughened surface with PureFix™ HA. The cup is available in a range of sizes and is indicated for primary and revision procedures.

A standard operative technique will be employed by all study surgeons, using the posterior approach. The routine post-operative patient care protocol of the study centre will be employed.

10 year implant survival is the primary aim, but in addition functional and radiographical outcome will be assessed a 1, 2, 5, 7 and 10 years.

ELIGIBILITY:
Inclusion Criteria:

1. Patients undergoing planned primary total hip arthroplasty with standard implants, suitable for the use of the uncemented Trident® II acetabular component.
2. Patients aged 18-75
3. Patients willing and able to comply with the study protocol
4. Patients that provide informed consent

Exclusion Criteria:

1. Patients not meeting study inclusion criteria
2. Bone stock that is inadequate for support or fixation of the prosthesis
3. Patients with a body mass index (kg/m2) >40
4. Procedures performed for pain relief in those with severely restricted mobility

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 125 (Estimated)
Dates: Start 2022-06-01 (Actual); Primary Completion 2024-11-25 (Actual); Study Completion 2034-11-25 (Estimated)

PRIMARY OUTCOMES:
Implant survival | 10 years
  All failures or revision of the Trident® II components as well as liner revisions will be documented.

SECONDARY OUTCOMES:
Oxford hip score | Preoperative, 1, 2, 5, 7 and 10 years
  The Oxford Hip Score is a patient reported outcome measure that was developed specifically to measure the impact of pain and functional disability in patients undergoing hip replacement. It consists of 12-questions and is scored using a 5-item Likert response format, reported on a 0 (worst) to 48 (best) scale with higher scores representing better outcomes. It is an extensively validated and widely adopted outcome measure in patients undergoing hip replacement surgery.
Forgotten Joint Score | Preoperative, 1, 2, 5, 7 and 10 years
  The Forgotten Joint Score-12 is a patient-reported outcome scale to assess joint awareness in hips during various activities of daily living. It uses a 5-point Likert response format, consists of 12-questions and the raw score is transformed to range from 0 (worst) to 100 (best) points. High scores indicate good outcome, i.e. a high degree of being able to forget about the affected joint in daily life. The FJS has a low ceiling effect and especially discriminates between good, very good and excellent outcome after THA and TKA. In its validation study it showed high internal consistency and discriminated well between patient groups known to show different outcome.
Short Form 12 | Preoperative, 1, 2, 5, 7 and 10 years
  The Short Form 12 is a 12-item questionnaire used to assess generic health outcomes from the patient's perspective. The SF-12 results in two summary scores: the physical and mental components summary (PCS and MCS) scores. This score is calculated using norm-based methodology and population mean scores. Both PCS and MCS have a population mean score of 50 with an standard deviation of 10.
EuroQol 5-dimension | Preoperative, 1, 2, 5, 7 and 10 years
  The EuroQol 5-dimension is a standardised instrument with five items for use as a measure of self-reported general health. Applicable to a wide range of health conditions and treatments, it provides a simple descriptive profile and a single index value for health status. This index for the UK population is on a scale of -0.594 to 1, where 1 represents perfect health and 0 represents death, with a utility of less than 0 being worse than death. It is one of the most frequently used measures to gain quality of life scores for analysis in health economy as utility weights for calculating quality of life adjusted life years (QALYs) can be obtained
Hip pain | Preoperative, 1, 2, 5, 7 and 10 years
  Global hip pain severity will be assessed using an 11 point (0-10) numerical rating scale (NRS), where 0 represents no pain and 10 the worst possible pain. The validity and sensitivity of the NRS has been well documented. As it has been suggested that using multiple measurements of pain status as opposed to a single value of 'current pain' may provide more realistic and meaningful measurements of pain intensity, separate assessments will be made of 'worst pain' and 'perceived mean daily pain' as has been specifically recommended for use in OA clinical trials.
Patient satisfaction | Preoperative, 1, 2, 5, 7 and 10 years
  Satisfaction questions are reported using a 5-point Likert response format hip (very satisfied, satisfied, unsure, dissatisfied or very dissatisfied). Specifically, questions will ask patients as to their
  1. overall satisfaction with their operated hip
  2. how well the surgery relieves pain in the operated joint
  3. how well surgery increases the ability to perform regular activities of daily living and to perform heavy work or sport activities
Radiographic (x-ray) assessment | Preoperatively, 1, 5 and 10 years
  Plain radiographs will be obtained for assessment of fixation of the device evaluating radiolucent lines (mm), cup abduction angle (degrees), anteversion (degrees) and cup-centre-edge angle (degrees). Plain radiographs will be divided into the three acetabular zones according to those defined by DeLee and Charnley. Radiolucent lines will be defined as less then 2mm, more than this will be defined a lysis. Lysis in all three acetabular zone will define a loose cup. Acetabular component inclination and version will be calculated from anteroposterior radiographs of the hip and/or hip and pelvis using established and validated techniques. The safe zones for acetabular component positioning were assessed using the commonly adopted parameters defined by Lewinnek et al. (inclination of 30° to 50° and anteversion of 5° to 25°) and Callanan et al. (inclination of 30° to 45° and anteversion of 5° to 25°).

CONTACTS AND LOCATIONS:
Overall Officials: Paul Gaston, MBChB, FRCS, Principal Investigator — NHS Lothian
Locations (1):
- NHS Lothian, Edinburgh, Lothian, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Due to patient confidentiality there is no plans to share patient level data.

REFERENCES:
- [Background] Dawson J, Fitzpatrick R, Carr A, Murray D. Questionnaire on the perceptions of patients about total hip replacement. J Bone Joint Surg Br. 1996 Mar;78(2):185-90. PMID 8666621
- [Background] Behrend H, Giesinger K, Giesinger JM, Kuster MS. The "forgotten joint" as the ultimate goal in joint arthroplasty: validation of a new patient-reported outcome measure. J Arthroplasty. 2012 Mar;27(3):430-436.e1. doi: 10.1016/j.arth.2011.06.035. Epub 2011 Oct 13. PMID 22000572
- [Background] Ware J Jr, Kosinski M, Keller SD. A 12-Item Short-Form Health Survey: construction of scales and preliminary tests of reliability and validity. Med Care. 1996 Mar;34(3):220-33. doi: 10.1097/00005650-199603000-00003. PMID 8628042
- [Background] EuroQol Group. EuroQol--a new facility for the measurement of health-related quality of life. Health Policy. 1990 Dec;16(3):199-208. doi: 10.1016/0168-8510(90)90421-9. PMID 10109801
- [Background] DeLee JG, Charnley J. Radiological demarcation of cemented sockets in total hip replacement. Clin Orthop Relat Res. 1976 Nov-Dec;(121):20-32. PMID 991504
- [Background] Liaw CK, Hou SM, Yang RS, Wu TY, Fuh CS. A new tool for measuring cup orientation in total hip arthroplasties from plain radiographs. Clin Orthop Relat Res. 2006 Oct;451:134-9. doi: 10.1097/01.blo.0000223988.41776.fa. PMID 16721351
- [Background] Park YS, Shin WC, Lee SM, Kwak SH, Bae JY, Suh KT. The best method for evaluating anteversion of the acetabular component after total hip arthroplasty on plain radiographs. J Orthop Surg Res. 2018 Apr 2;13(1):66. doi: 10.1186/s13018-018-0767-4. PMID 29609639
- [Background] Lewinnek GE, Lewis JL, Tarr R, Compere CL, Zimmerman JR. Dislocations after total hip-replacement arthroplasties. J Bone Joint Surg Am. 1978 Mar;60(2):217-20. PMID 641088
- [Background] Callanan MC, Jarrett B, Bragdon CR, Zurakowski D, Rubash HE, Freiberg AA, Malchau H. The John Charnley Award: risk factors for cup malpositioning: quality improvement through a joint registry at a tertiary hospital. Clin Orthop Relat Res. 2011 Feb;469(2):319-29. doi: 10.1007/s11999-010-1487-1. PMID 20717858
- See also: Edinburgh Orthopaedic home page — https://www.edinburghorthopaedics.org/